CLINICAL TRIAL: NCT05815953
Title: The Polarstem Versus Corail; a Comparison of Micromotion and Periprosthetic Bone Remodelling of Two Femoral Stems. A Randomised Trial of 60 Patients Using Radiostereometric Analysis, Dual Energy X-ray Absorptiometry and Computer Tomography
Brief Title: Polarstem Versus Corail; a Comparison of Micromotion and Periprosthetic Bone Remodelling of Two Femoral Stems
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse-Bergen HF (Other)
Collaborators: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Principal Investigator, Geir Hallan, Clinical Professor, Helse-Bergen HF
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27379
Record Dates: First submitted 2022-04-29; First posted 2023-04-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Arthritis of the Hip
Keywords: Arthroplasty, Replacement; Arthroplasty, Replacement, Hip; Osteoarthritis; Osteoarthritis, Hip; Arthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip; Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Computer generated block randomization for each participating surgeon. The envelopes are sequentially numbered, opaque and sealed. The surgeon is not blinded, but the patient and the physiotherapist that do the clinical follow-ups are.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polarstem (Experimental): Polarstem uncemented femoral stem
  Interventions: Device: Polarstem
- Corail (Active Comparator): Corail uncemented femoral stem
  Interventions: Device: Corail

INTERVENTIONS:
Device: Polarstem — Stem used in total hip replacement. Manufacturer: Smith & Nephew Orthopaedics AG, Baar, Switzerland.
  Arms: Polarstem
Device: Corail — Stem used in total hip replacement. Manufacturer: De Puy Int Ltd, Leeds, UK.
  Arms: Corail

SUMMARY:
A randomised controlled trial comparing a recently introduced femoral stem with an established stem for total hip arthroplasty (THA). 60 patients will be randomised into one of the two groups

1. Polarstem uncemented femoral stem (Smith & Nephew)
2. Corail uncemented femoral stem (De Puy) All patients will receive a 32mm cobalt-chromium (CoCr) femoral head and an R3 acetabular cup with a 10 Mrad highly cross-linked polyethylene (XLPE) liner (Smith & Nephew).

Radiostereometric analysis (RSA) will be used to measure stem migration. Dual-energy x-ray absorptiometry (DXA) measurements will be used to measure bone mineral density. Clinical outcome will be assessed at different time point to evaluate satisfaction and function. Data from the Norwegian Arthroplasty Register will be used to investigate the risk of revision.

DETAILED DESCRIPTION:
The gold standard in THA the last 45 years has been the all-cemented metal-on polyethylene prostheses such as the Charnley low-frictional arthroplasty. From 1980 and onwards however, uncemented THA have been increasingly popular worldwide, especially for the younger patients. The reasons for this were reports on poor results of the Charnley cemented THA in young patients, and the belief that the cement itself was the cause of periprosthetic osteolysis and loosening of the prostheses. Uncemented THA have good results in some reports and poor results in others. The modern uncemented femoral stems have proven good or even excellent results at medium to long term follow-up in the register and in other clinical studies. The Corail uncemented femoral stem (DePuy) has dominated the Norwegian market on uncemented stems since the mid 1980'ies. Its clinical performance is well documented with good results in terms of implant survival5. The Polarstem (Smith & Nephew) was introduced in 2002 by a group of surgeons that believed the Corail stem had certain limitations, and the Polarstem is a Corail-like stem with some modifications. The basic design philosophy of a straight tapered design is the same for both stems.

Unlike drugs, medical devices such as orthopaedic implants can be launched on the market without any proof of clinical efficacy. In some cases, inferior implants have been used in thousands of patients before the inferior results were discovered. Some authors propose a stepwise introduction of new implants in order to avoid compromising large numbers of patients. The present study is a step in the introduction of a relatively new femoral stem. High accuracy measuring tools will be used to measure critical factors such as implant migration and bone remodelling at short-term follow-up. The findings will give information on the expected clinical outcome at longer term.

The aims of the study are

* To compare the migration of the Polarstem and the Corail stem with RSA. The null hypothesis is that there is no difference in the early (2 years postoperative) migration of these implants. Early migration has earlier proved to be a surrogate for implant performance at medium and long term.
* To compare any remodeling of periprosthetic femoral bone from direct postoperative measures to later time points. Periprosthetic bone loss, especially in the proximal femur, can compromise the longevity of a prosthetic joint. This bone loss vary and will be compared between the two designs.
* To assess and compare clinical outcome measures and radiological outcomes such as signs of loosening and osteolysis.

Components

* The Polarstem uncemented femoral stem (Smith & Nephew Orthopaedics AG, Baar, Switzerland) is a straight titanium alloy (Ti6Al4V), tapered, fully hydroxyapatite (HA) coated uncemented implant. HA is used to enhance on-growth of bone to the implant surface and is put on top of a plasma spray porous coating (titanium) in a 150 + 75µm layer. The stem was introduced onto the market in 2002, and no documentation on the clinical efficacy beyond 5 years existed when this study was planned. The design philosophy however is similar to other implants that have good results at long term.
* The Corail uncemented femoral stem (De Puy Int Ltd, Leeds, UK) is a straight, tapered fully hydroxyl-apatite coated stem that was introduced in 1986 in Norway. It has been the most commonly used uncemented stem since, and by 2014 more than 60% of THA patients in Norway received this stem. The 15 year survival was 97% according to a study from 2007.
* R3 uncemented acetabular cup (Smith & Nephew Orthopaedics AG, Baar, Switzerland) is a fourth-generation hemispheric, porous coated cup intended for press-fit fixation. The cup is based on the well-documented Reflection cup (also Smith & Nephew) and has a locking mechanism that has proved better stability of the liner in laboratory studies. Further, a new asymmetric coating made of titanium powder (StikTite) with higher porosity and friction has been added. The stability of this cup was found to be excellent in a series of patients measured by RSA. The R3 cup was approved by the European Commission (CE) in 2007 and the Food and Drug Administration (FDA) in 2008. In some countries such as Australia the implant is one of the most frequently used, and according to the Australian Orthopaedic Association National Joint Replacement Registry (AOANJRR) the results with up to 5 years of follow-up are promising.

Radiography

* Radiostereometric analysis (RSA) is a highly accurate and precise method of evaluating implant migration and polyethylene wear. The precision usually is about 0.1-0.4 mm (translational migration) and 0.1-1 degrees (rotation). The radiation dose is low compared to plain x-rays (10-20%). During surgery, tiny spheres of Tantalum are implanted in periprosthetic bone. The metal implants will be measured with markerless RSA. On day 1-6 postoperatively, two simultaneous exposures of the hip and a co-ordinate system are taken. These films allow three-dimensional definition of the implant and bone relative to the co-ordinate system. Implant migration and rotation is measured on repeat examinations over time. The high precision allows us to detect small differences between groups, and also means that the number of subjects in each group can be restricted. The precision (repeatability) of the measurements in this study will be evaluated by double examinations at the 1-year RSA-visit. Limits for significant differences are calculated as the 99% confidence intervals of the absolute mean values of the double examinations.
* Plain x-rays. At all follow-up consultations plain x-rays of the pelvis, and an AP and lateral view of the hip will be taken. On postoperative pelvic views the varus/valgus position of the stem, and cup inclination will be measured. Later these values will be evaluated together with migration- and wear values. Osteolysis will be measured.
* Computed tomography. In order to investigate the incidence and to quantify periprosthetic osteolysis investigators will perform CT scanning of the patients at 10 years.
* Dual x-ray absorptiometry (DXA). Periprosthetic femoral bone mineral density (BMD) will be measured with DXA. The load transmission to periprosthetic bone differs according to the mechanical properties and design of the implant. Stress-shielding (stress-protection) of periprosthetic bone results in local osteopenia, bone loss, and may contribute to loosening, periprosthetic fractures and complex revision procedures. Most contemporary hip implant designs aim to reduce stress shielding as much as possible.

Our department's standard surgical approach, the posterolateral approach, will be used on all patients. The operations will take place in an operation theatre with laminar airflow, the patients will receive prophylactic antibiotics (Cephalotin 2gx4, or Clindamycin 0.6gx3 if Penicillin allergy) perioperatively, and prophylactics against thromboembolism (Dalteparin 5000 international units for 2 weeks). Implantation of the prosthetic components will be done according to preoperative planning and the manufacturer's advice. 6-10 tantalum beads (Ø=1mm) will be inserted into the proximal femur. The holes are then covered with bone wax.

The patients are allowed immediate weight bearing as tolerated. Walking aids at demand. Physiotherapy is started on day 1 postoperatively and is continued at dismission.

The results of the RSA- and DXA-examinations and clinical outcome measures will be collected in electronic files under the respective patient numbers. Data obtained on previous occasions will not be accessible when examining the patient.

According to the Data Inspectorate, the requirements for a simple 'melding' are

* The responsible (medical doctor) investigator is employed by the organization in which the patient is being registered.
* The patient gives his/her written consent to participation in the study.
* The end of the study is determined at its start.
* The gathered data are deleted or anonymized at the end of the study.
* The study does not electronically merge data from different person registers.

These requirements are fulfilled in the present study, and a "melding" will be submitted to the Data Inspectorate when the administrative details concerning the study are ready.

A patient list will be made coupling patient name and personal identification number to a number on the patient list (1 through 60). The project leader is responsible for the safe handling of the list. Other forms with patient information are labelled with the patient number only for identification. The sponsors of the study will have access to the anonymised data. The study is reported to 'Personvernombudet' through 'Norsk samfunnsvitenskapelig datatjeneste i Bergen'.

Analysis of variance on repeated measurements (ANOVA) will be used on the RSA- and on the clinical data if the data are normally distributed. In our earlier RSA studies, the data have displayed normal distribution. If however, the data are not normally distributed, non-parametric tests (Mann-Whitney U-test, Wilcoxon matched-pairs test) will be used.

Adverse effects, side effects, and unfortunate effects of the surgery will immediately be reported to the project leader and to the sponsors. Abortion or abruption of the study will be considered in the case of unexpected complications.

Funding will be applied for from:

* The Regional Health Services (Helse Vest Regionale helseforetak, Det regionale samarbeidsorganet, Helse Bergen, Haukeland Universitetssykehus, 5021 BERGEN, Norway)
* Smith & Nephew Orthopaedics AG, Baar, Switzerland

The study will be performed at the Department of Orthopaedic Surgery, Haukeland University Hospital, Bergen, Norway.

ELIGIBILITY:
Inclusion Criteria:

* primary arthritis
* secondary arthritis
* aseptic necrosis of the femoral head
* acute hip fracture
* sequelae after hip fracture
* can use standard implants

Exclusion Criteria:

* active malignant disease
* rheumatoid arthritis or other generalised auto-immune arthritic disease
* BMI>35
* insulin dependent diabetes mellitus
* chronic or recurrent infection
* liver disease
* Pagets disease
* dementia or lack of compliance for other reasons
* uncompensated cardiac- or pulmonary disease (ASA class 3 or 4)

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2033-01-31 (Estimated)

PRIMARY OUTCOMES:
Migration of femoral component into the bone; Change from baseline to the prescribed time | Baseline (1, 2 or 3 days after operation; post-operative), 3 months, 12 months, 24 months, 60 months, and 10 years postoperatively.
  Radiostereometric pictures will be taken within 1, 2 or 3 days after operation (post-operative) to have a baseline and at the prescribed intervals.
  Migration will be measure with radiostereometric analysis (RSA) at the described intervals. Implant migration the first few years after implantation can correspond to loosening at long term.
Periprosthetic femoral bone mineral density (BMD); Change from baseline (postoperative) to the prescribed time | Baseline (1, 2 or 3 days after operation; post-operative), 24 months and 60 months after surgery.
  Periprosthetic femoral bone mineral density (BMD) will be measured within 1, 2 or 3 days after operation (post-operative) to have a baseline and at the prescribed intervals using Dual x-ray absorptiometry (DXA). A DXA-machine (Lunar Prodigy, GE) located at the Department of Rheumatology at Haukeland University Hospital will be used with customized software.

SECONDARY OUTCOMES:
Harris Hip Score (HHS); Change from pre-operative to the prescribed time | Pre-operative, 3 months, 12 months , 24 months, 60 months, and 10 years after surgery.
  Clinical reported outcome. HHS was designed to be a standardized assessment of patients following total hip arthroplasty. Since that time, it has also been used for evaluating patients following hip fractures and the diagnosis of osteoarthritis.
  The HHS is a physician-completed instrument that consists of subscales for pain severity (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 0-4 points), and range of motion (2 items, 0-5 points). Scores range from 0 (worse disability) to 100 (less disability).(Obtained from Free online Harris Hip score calculator - OrthoToolKit, red 06.01.2021)
Hip Disability and Osteoarthritis Outcome Score (HOOS); Change from pre-operative to the prescribed time | Pre-operative, 3 months, 12 months , 24 months, 60 months, and 10 years after surgery.
  Patient reported outcome. HOOS assesses patient pain (10 items), satisfaction including stiffness and range of motion (5 items), activity limitations-daily living (17 items), sports and recreation function (4 items), and hip related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible hip symptoms and 100 indicating no hip symptoms. This is a patient reported joint-specific score, which may be useful for assessing changes in hip pathology over time, with or without treatment (obtained from Free online HOOS score calculator - OrthoToolKit, red 06.01.2021)
EQ-5D-3L; Change from pre-operative to the prescribed time | Pre-operative, 3 months, 12 months , 24 months, 60 months, and 10 years after surgery.
  Patient reported outcome. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. (Obtained from https://euroqol.org/eq-5d-instruments/eq-5d-3l-about/, red 06.01.2021)
EQ VAS; Change from pre-operative to the prescribed time | Pre-operative, 3 months, 12 months , 24 months, 60 months, and 10 years after surgery.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement. (Obtained from https://euroqol.org/eq-5d-instruments/eq-5d-3l-about/, red 06.01.2021)
Hip pain; Change from pre-operative to the prescribed time | Pre-operative, 3 months, 12 months , 24 months, 60 months, and 10 years after surgery.
  Patient reported outcome using Visual Analogue Scale (VAS) from 0-100 0 is no pain, 100 is worst imaginable pain.
Satisfaction with the Hip; Change from pre-operative to the prescribed time | Pre-operative, 3 months, 12 months , 24 months, 60 months, and 10 years after surgery.
  Patient reported outcome using Likert scale from 1-5. 1 is very satisfied, 5 is very litle satisfied
Position of the stem: Varus/valgus | Baseline (1, 2 or 3 days after operation; post-operative)
  Pelvic views from x-ray will be used to measure varus/ valgus
Position of the stem: Cup inclination | Baseline (1, 2 or 3 days after operation; post-operative)
  Pelvic views from x-ray will be used to measure cup inclination
Position of the stem; Change from baseline to the prescribed time | Baseline (1, 2 or 3 days after operation; post-operative), 12 months, 24 months, 60 months, and 10 years postoperatively.
  Implant positioning parameters (inclination, version, offset) are measured useing anterior-posterion and plain radiographs
Osteolysis in Acetabulum; Change from baseline to the prescribed time | Baseline (1, 2 or 3 days after operation; post-operative), 12 months, 24 months, 60 months, and 10 years postoperatively.
  Anterior-posterior x-ray will be taken and based on this Osteolysis in acetabulum will be classified using Paproskys classification (type I, IIA, IIB, IIC, IIIA, IIIB).
Osteolysis in Femur; Change from baseline to the prescribed time | Baseline (1, 2 or 3 days after operation; post-operative), 12 months, 24 months, 60 months, and 10 years postoperatively.
  Anterior-posterior x-ray will be taken and based on this Osteolysis in femur will be classified using Paproskys classification (type I, II, IIIA, IIIB, IV).

CONTACTS AND LOCATIONS:
Overall Officials: Geir Hallan, MD; PhD, Study Director — Department of Orthopaedic Surgery, Haukeland University Hospital, Bergen, Norway; Ove N Furnes, MD; PhD, Study Chair — Department of Orthopaedic Surgery, Haukeland University Hospital, Bergen, Norway; Torbjørn B Kristensen, MD; PhD, Study Chair — Department of Orthopaedic Surgery, Haukeland University Hospital, Bergen, Norway; Jan-Erik Gjertsen, MD; PhD, Study Chair — Department of Orthopaedic Surgery, Haukeland University Hospital, Bergen, Norway; Paul J Høl, PhD, Study Chair — Department of Orthopaedic Surgery, Haukeland University Hospital, Bergen, Norway; Irene O Moldestad, MSc, Study Chair — Department of Orthopaedic Surgery, Haukeland University Hospital, Bergen, Norway
Locations (1):
- Helse Bergen HF, Bergen, Postbox 1400, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandler HP, Reineck FT, Wixson RL, McCarthy JC. Total hip replacement in patients younger than thirty years old. A five-year follow-up study. J Bone Joint Surg Am. 1981 Dec;63(9):1426-34. No abstract available. PMID 7320033
- [Background] Carlsson AS, Gentz CF. Mechanical loosening of the femoral head prosthesis in the Charnley total hip arthroplasty. Clin Orthop Relat Res. 1980 Mar-Apr;(147):262-70. PMID 7371307
- [Background] Jones LC, Hungerford DS. Cement disease. Clin Orthop Relat Res. 1987 Dec;(225):192-206. PMID 3315375
- [Background] Vervest TM, Anderson PG, Van Hout F, Wapstra FH, Louwerse RT, Koetsier JW. Ten to twelve-year results with the Zweymuller cementless total hip prosthesis. J Arthroplasty. 2005 Apr;20(3):362-8. doi: 10.1016/j.arth.2004.11.017. PMID 15809956
- [Background] Hallan G, Lie SA, Furnes O, Engesaeter LB, Vollset SE, Havelin LI. Medium- and long-term performance of 11,516 uncemented primary femoral stems from the Norwegian arthroplasty register. J Bone Joint Surg Br. 2007 Dec;89(12):1574-80. doi: 10.1302/0301-620X.89B12.18969. PMID 18057355
- [Background] Parvizi J, Keisu KS, Hozack WJ, Sharkey PF, Rothman RH. Primary total hip arthroplasty with an uncemented femoral component: a long-term study of the Taperloc stem. J Arthroplasty. 2004 Feb;19(2):151-6. doi: 10.1016/j.arth.2003.10.003. PMID 14973856
- [Background] Soderman P, Malchau H. Is the Harris hip score system useful to study the outcome of total hip replacement? Clin Orthop Relat Res. 2001 Mar;(384):189-97. doi: 10.1097/00003086-200103000-00022. PMID 11249165
- [Background] Karrholm J, Borssen B, Lowenhielm G, Snorrason F. Does early micromotion of femoral stem prostheses matter? 4-7-year stereoradiographic follow-up of 84 cemented prostheses. J Bone Joint Surg Br. 1994 Nov;76(6):912-7. PMID 7983118
- [Background] Valstar ER, Gill R, Ryd L, Flivik G, Borlin N, Karrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthop. 2005 Aug;76(4):563-72. doi: 10.1080/17453670510041574. PMID 16195075
- [Background] Harris WH. Traumatic arthritis of the hip after dislocation and acetabular fractures: treatment by mold arthroplasty. An end-result study using a new method of result evaluation. J Bone Joint Surg Am. 1969 Jun;51(4):737-55. No abstract available. PMID 5783851
- [Background] Karrholm J, Herberts P, Hultmark P, Malchau H, Nivbrant B, Thanner J. Radiostereometry of hip prostheses. Review of methodology and clinical results. Clin Orthop Relat Res. 1997 Nov;(344):94-110. PMID 9372762
- [Background] Mirsky EC, Einhorn TA. Bone densitometry in orthopaedic practice. J Bone Joint Surg Am. 1998 Nov;80(11):1687-98. doi: 10.2106/00004623-199811000-00018. No abstract available. PMID 9840640
- [Background] Bourne RB, McCalden RW, Naudie D, Charron KD, Yuan X, Holdsworth DW. The next generation of acetabular shell design and bearing surfaces. Orthopedics. 2008 Dec;31(12 Suppl 2):orthosupersite.com/view.asp?rID=37179. PMID 19298027
- See also: Australian Orthopaedic Association National Joint Replacement Registry. Annual report 2015 — https://aoanjrr.sahmri.com/documents/10180/217745/Hip+and+Knee+Arthroplasty
- See also: Malchau, Henrik 1995, Doctoral Theses: "On the importance of stepwise introduction of new hip implant technology : assessment of total hip replacement using clinical evaluation, radiostereometry, digitised radiography and a national hip registry" — http://hdl.handle.net/2077/12932